CLINICAL TRIAL: NCT03703739
Title: Effect of Solubilizing Agents on Iron Absorption From Iron Fortified Rice in Young Women
Brief Title: Iron Absorption From Iron Fortified Extruded Rice Co-fortified With Various Solubilizing Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Iron_RiceSolubilizing
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Iron-deficiency
Keywords: Iron deficiency; iron fortified rice; extruded rice
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Reference meal 1 (Active Comparator): 50 g of Commercial Rice (Jasmin Rice) (dry weight) was cooked and 4 mg iron from Ferrous sulfate was added Prior to give to participants. Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Reference meal 1
- Reference 2 (Active Comparator): 50 g of Commercial Rice (Jasmin Rice) (dry weight) was cooked and 4 mg iron from Ferrous sulfate was added Prior to give to participants. Rice meal consumed with bean sauce.
  Interventions: Dietary Supplement: Reference 2
- Test meal A (Experimental): Commercial Rice (Jasmin Rice) was mixed with iron fortified extuded rice cofortified with zinc oxide and ethylenediaminetetraacetic acid (mixing ratio 100:1), Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal A
- Test meal B (Experimental): Commercial Rice (Jasmin Rice) was mixed with iron fortified extuded rice co-fortified with zinc sulfate and ethylenediaminetetraacetic acid (mixing ratio 100:1), Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal B
- Test meal C (Experimental): Commercial Rice (Jasmin Rice) was mixed with iron fortified extuded rice co-fortified with zinc sulfate, citric acid and trisodium citrate (mixing ratio 100:1), Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal C
- Test meal D (Experimental): Commercial Rice (Jasmin Rice) was mixed with iron fortified extuded rice co-fortified with zinc sulfafe and sodium pyrophosphate (mixing ratio 100:1), Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal D
- Test meal E (Experimental): Commercial Rice (Jasmin Rice) was mixed with iron fortified extuded rice co-fortified with zinc sulfate, citric acid and trisodium citrate (mixing ratio 100:1), Rice meal consumed with bean Sauce.
  Interventions: Dietary Supplement: Test meal E

INTERVENTIONS:
Dietary Supplement: Reference meal 1 — 1 ml Ferrous sulfate solution (4mgFe/ml) was added in cooked comercial Rice Prior to served to participant. The meal served with 30 g mixed vegetable Sauce and 300 ml nanopure water
  Arms: Reference meal 1
Dietary Supplement: Reference 2 — 1 ml Ferrous sulphate solution (4mgFe/ml) was added in cooked comercial Rice Prior to served to participant. The meal served with 30 g bean Sauce and 300 ml nanopure water
  Arms: Reference 2
Dietary Supplement: Test meal A — Fortified extruded Rice was mixed with Commercial Rice (mixing Ratio: 1:100) The meal served with 30 g vegetable Sauce and 300 ml nanopure water.
  ** composition of extruded Rice: Ferric pyrophosphate, zinc oxide and ethylenediaminetetraacetic acid
  Arms: Test meal A
Dietary Supplement: Test meal B — Fortified extruded Rice was mixed with Commercial Rice (mixing Ratio: 1:100) The meal served with 30 g vegetable Sauce and 300 ml nanopure water.
  ** composition of extruded Rice: Ferric pyrophosphate, zinc sulfate and ethylenediaminetetraacetic acid
  Arms: Test meal B
Dietary Supplement: Test meal C — Fortified extruded Rice was mixed with Commercial Rice (mixing Ratio: 1:100) The meal served with 30 g vegetable Sauce and 300 ml nanopure water.
  ** composition of extruded Rice: Ferric pyrophosphate, zinc sulfate, citric acid and trisodium Citrate.
  Arms: Test meal C
Dietary Supplement: Test meal D — Fortified extruded Rice was mixed with Commercial Rice (mixing Ratio: 1:100) The meal served with 30 g vegetable Sauce and 300 ml nanopure water.
  ** composition of extruded Rice: Ferric pyrophosphate, zinc sulfate and sodium pyrophosphate.
  Arms: Test meal D
Dietary Supplement: Test meal E — Fortified extruded Rice was mixed with Commercial Rice (mixing Ratio: 1:100) The meal served with 30 g bean Sauce and 300 ml nanopure water.
  ** composition of extruded Rice: Ferric pyrophosphate, zinc sulfate, citric acid and trisodium Citrate.
  Arms: Test meal E

SUMMARY:
Food fortification is regarded as a safe and cost-effective approach to counteract and prevent iron deficiency. Rice is a staple food for millions of people living in regions where iron-deficiency anaemia is a significant public health problem. Therefore, rice may be a promising fortification vehicle. Ferric pyrophosphate (FePP) is an acceptable iron compound for rice fortification, due to its white colour and low reactivity with the rice matrix. However, iron from FePP generally has a low bioavailability. To increase the low iron bioavailability of FePP in fortified rice, ligands acting as solubilizing agents have been suggested, such as citric acid/trisodium citrate (CA/TSC), ethylenediaminetetraacetic acid (EDTA) and sodium pyrophosphate (NaPP).

It is however unclear to which extent CA/TSC would enhance iron bioavailability in presence of phytic acid, a common inhibitor of iron absorption found in whole grains and legumes. Zinc oxide reduces iron bioavailability from FePP with and without CA/TSC, in contrast to Zinc sulphate. It is however unclear if this decrease would be also expected in presence of EDTA as solubilizing agent. Further, NaPP has been suggested as a solubilizing agent, enhancing the bioavailability from FePP in bouillon cubes. This study aim to test its effect in rice. Meals containing a high (bean sauce) and low (mixed vegetable) phytic acid level sauce will be used to simulated varying dietary backgrounds, allowing to answer the question which solubilizing agent is viable in enhancing iron bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 40 years old
* Normal body Mass Index (18.5 - 25 kg/m2)
* Body weight ≤ 65 kg
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by self-declaration)
* Lactating up to 6 weeks before study initiation
* Anaemia (Hb < 12.0 g/dL)
* Elevate CRP (>5.0 mg/L)
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using Fe stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol (e.g. not available on certain study appointments)
* Smokers (> 1 cigarette per week)
* Difficulties with blood sampling
* Male gender
* Do not understand English

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 2 in the isotopic ratio of iron in blood at week 4 | 2 weeks, 4 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 4 in the isotopic ratio of iron in blood at week 6 | 4 weeks, 6 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 6 in the isotopic ratio of iron in blood at week 8 | 6 weeks, 8 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 8 in the isotopic ratio of iron in blood at week 10 | 8 weeks, 10 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.

SECONDARY OUTCOMES:
Haemoglobin | 2, 4,6,8 and 10 weeks
  Haemoglobin of each timepoint
Plasma Ferritin | 2, 4, 6, 8 and 10 weeks
  Plasma Ferritin of each timepoint
Inflammation Marker | 2, 4, 6, 8 and 10 weeks
  Plasma Ferririn of each timepoint

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Scheuchzer P, Syryamina VN, Zimmermann MB, Zeder C, Nystrom L, Yulikov M, Moretti D. Ferric Pyrophosphate Forms Soluble Iron Coordination Complexes with Zinc Compounds and Solubilizing Agents in Extruded Rice and Predicts Increased Iron Solubility and Bioavailability in Young Women. J Nutr. 2023 Mar;153(3):636-644. doi: 10.1016/j.tjnut.2022.12.003. Epub 2022 Dec 24. PMID 36931746